CLINICAL TRIAL: NCT05751694
Title: Effectiveness of Visceral Manual Therapy in Bruxist Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Lourdes María Fernández Seguín, Assistant Professor. Physiotherapy Department, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 070223TDCNR
Record Dates: First submitted 2023-02-08; First posted 2023-03-02 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-05

CONDITIONS: Bruxism
Keywords: Bruxism; Musculoskeletal Manipulations; Physical Therapy Modalities; Autonomic Nervous System
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visceral manual treatment (Experimental): The objective of this technique is to reduce the tension of the tissues of the epigastric area.
  Interventions: Procedure: Visceral manual treatment
- Respiratory listening (Active Comparator): It is a maneuver to evaluate the mobility of the ribs during respiration.
  Interventions: Procedure: Respiratory listening

INTERVENTIONS:
Procedure: Visceral manual treatment — The patient will be placed in a reclining sitting position and triple flexion of the lower limbs to keep the abdominal region relaxed. The therapist will be placed to the right of the patient at the height of the abdomen, with the hands placed in the epigastric area. He will make a skin fold that reduces tension in the area, so that the contact is focused on the visceral tissue of the area. The patient will be asked to take deep breaths, and during the exhalation, the therapist will perform a zigzag movement with vibration of the hands while pulling the tissue caudally. This procedure will be performed for 5 minutes.
  Arms: Visceral manual treatment
Procedure: Respiratory listening — The patient and the therapist will be placed in the same position as in the experimental group. The therapist will place his hands in contact with the lower rib cage, and the patient will be asked to take a deep breath. The therapist will not exert any pressure, nor place restrictions on the tissues or movements of the ribcage.
  Arms: Respiratory listening

SUMMARY:
Objective: check the effectiveness of visceral manual therapy on bruxist patients Design: Experimental, analytical, longitudinal, prospective, randomized, single-blind study with a blinded evaluator.

Subjects: 68 subjects over 18 years old, with bruxism (diagnoses by a dentist). Methods: Subjects will be randomized into 2 groups: an experimental group (EG) to which a visceral manual technique will be applied and a control group (CG) to which a placebo manual technique will be administered. Both groups will receive 2 interventions one week apart. The measurements will be made before and after the interventions, and a last measurement will be made one month after the last intervention. Therefore, the patient will visit the center 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with bruxism diagnosed and referred by a dentist
* Age: older than 18 years-old.

Exclusion Criteria:

* Recent craniofacial, mandibular or cervical trauma or fracture.
* Temporomandibular joint surgery.
* Acute pain due to other components of the masticatory system (caries, inflammation of the dental root).
* Abdominal surgery.
* Gastric ulcers.
* Gastritis.
* Previous or current gastric neoplasm.
* Neurological or systemic diseases.
* Pregnant, including the period of breastfeeding.
* Patients receiving chemotherapy or radiotherapy.
* Cognitive, psychosomatic or psychiatric illnesses that may affect the data obtained.
* Basic systemic disease of rheumatic origin (for example, arthritis, osteoarthritis, gout and psoriasis).
* Cerebrovascular and brain diseases.
* Arrhythmia and other cardiac problems.
* Implanted electronic devices.
* Drug or alcohol abuse, analgesic or sedative therapy, and use of medications that affect the central nervous system (for example, antidepressants, anxiolytics, and anticonvulsants).
* Patients who have previous experience with manual treatment of the diaphragm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) Baseline-1 | Baseline pre-intervention
  The pressure pain threshold of the fourth cervical vertebra and masseter and temporal muscles will be evaluated using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
PPT Change-1 | Change from "PTT Baseline-1" immediately post-intervention
  The pressure pain threshold of the fourth cervical vertebra and masseter and temporal muscles will be evaluated using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
PPT Baseline-2 | Baseline pre-intervention at 7 days
  The pressure pain threshold of the fourth cervical vertebra and masseter and temporal muscles will be evaluated using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
PPT Change-2 | Change from "PTT Baseline-2" immediately post-intervention
  The pressure pain threshold of the fourth cervical vertebra and masseter and temporal muscles will be evaluated using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
PPT Change-3 | Change from "PTT Baseline-2" and "PTT Change-2" at 1 month
  The pressure pain threshold of the fourth cervical vertebra and masseter and temporal muscles will be evaluated using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Heart Rate Variability (HRV) Baseline-1 | Baseline pre-intervention
  Heart rate variability (HRV) was measured using a Polar H10 strap and the EliteHRV mobile app to collect the data. These data were exported to Kubios software to obtain HRV results. A 5-minute measurement was performed with the patient in the supine position.
HRV Change-1 | Change from "HRV baseline-1" inmediately post-intervention
  Heart rate variability (HRV) was measured using a Polar H10 strap and the EliteHRV mobile app to collect the data. These data were exported to Kubios software to obtain HRV results. A 5-minute measurement was performed with the patient in the supine position.
HRV Baseline-2 | Baseline pre-intervention at 7 days
  Heart rate variability (HRV) was measured using a Polar H10 strap and the EliteHRV mobile app to collect the data. These data were exported to Kubios software to obtain HRV results. A 5-minute measurement was performed with the patient in the supine position.
HRV Change-2 | Change from "HRV baseline-2" inmediately post-intervention
  Heart rate variability (HRV) was measured using a Polar H10 strap and the EliteHRV mobile app to collect the data. These data were exported to Kubios software to obtain HRV results. A 5-minute measurement was performed with the patient in the supine position.
HRV Change-3 | Change from "HRV baseline-2" and "HRV change-2" at 1 month
  Heart rate variability (HRV) was measured using a Polar H10 strap and the EliteHRV mobile app to collect the data. These data were exported to Kubios software to obtain HRV results. A 5-minute measurement was performed with the patient in the supine position.
Myotonometry baseline-1 | Baseline pre-intervention
  The muscle tone of the masseter muscle was assessed using a myotonometer (Myoton muscle diagnostics). 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Myotonometry change-1 | Change from "myotonometry baseline-1" inmediately post-intervention
  The muscle tone of the masseter muscle was assessed using a myotonometer (Myoton muscle diagnostics). 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Myotonometry baseline-2 | Baseline pre-intervention at 7 days
  The muscle tone of the masseter muscle was assessed using a myotonometer (Myoton muscle diagnostics). 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Myotonometry change-2 | Change from "myotonometry baseline-2" inmediately post-intervention
  The muscle tone of the masseter muscle was assessed using a myotonometer (Myoton muscle diagnostics). 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Myotonometry change-3 | Change from "myotonometry baseline-2" and "myotonometry change-2" at 1 month
  The muscle tone of the masseter muscle was assessed using a myotonometer (Myoton muscle diagnostics). 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.

SECONDARY OUTCOMES:
Cervical Range of Motion (CROM) Baseline-1 | Baseline pre-intervention
  The evaluator will place the CROM-device® goniometer on the patient's head. It will ask you for movements of flexion, extension, right and left side flexion, and right and left rotation of the cervical spine. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Cervical Range of Motion (CROM) Change-1 | Change from "CROM Baseline-1" immediately post-intervention
  The evaluator will place the CROM-device® goniometer on the patient's head. It will ask you for movements of flexion, extension, right and left side flexion, and right and left rotation of the cervical spine. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Cervical Range of Motion (CROM) Baseline-2 | Baseline pre-intervention at 7 days
  The evaluator will place the CROM-device® goniometer on the patient's head. It will ask you for movements of flexion, extension, right and left side flexion, and right and left rotation of the cervical spine. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Cervical Range of Motion (CROM) Change-2 | Change from "CROM Baseline-2" immediately post-intervention
  The evaluator will place the CROM-device® goniometer on the patient's head. It will ask you for movements of flexion, extension, right and left side flexion, and right and left rotation of the cervical spine. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Cervical Range of Motion (CROM) Change-3 | Change from "CROM Baseline-2" and "CROM Change-2" at 1 month
  The evaluator will place the CROM-device® goniometer on the patient's head. It will ask you for movements of flexion, extension, right and left side flexion, and right and left rotation of the cervical spine. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Perceived Stress Scale (PSS-14) Baseline | Baseline
  Perceived Stress Scale evaluates the level of perceived stress during the last month and consists of 14 items. The maximum score is 56 points. A higher score corresponds to a higher level of perceived stress.
PSS-14 Change | Change from Baseline PSS-14 at 1 month
  Perceived Stress Scale evaluates the level of perceived stress during the last month and consists of 14 items. The maximum score is 56 points. A higher score corresponds to a higher level of perceived stress.
Mandibular Mobility Baseline-1 | Baseline pre-intervention
  For the measurement of vertical opening and lateral deviation of the mandible, the TheraBite® range of motion™ will be used. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Mandibular Mobility Change-1 | Change from "Mandibular Mobility Baseline-1" immediately post-intervention
  For the measurement of vertical opening and lateral deviation of the mandible, the TheraBite® range of motion™ will be used. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Mandibular Mobility Baseline-2 | Baseline pre-intervention at 7 days
  For the measurement of vertical opening and lateral deviation of the mandible, the TheraBite® range of motion™ will be used. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Mandibular Mobility Change-2 | Change from "Mandibular Mobility Baseline-2" immediately post-intervention
  For the measurement of vertical opening and lateral deviation of the mandible, the TheraBite® range of motion™ will be used. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Mandibular Mobility Change-3 | Change from "Mandibular Mobility Baseline-2" and "Mandibular Mobility Change-2" at 1 month
  For the measurement of vertical opening and lateral deviation of the mandible, the TheraBite® range of motion™ will be used. 3 measurements will be made with a period of 30 seconds between measurements and we will obtain the average of the 3.
Pittsburgh Sleep Quality Index (PSQI) Baseline | Baseline
  It is a tool used to assess the quality of sleep in the last month.It consists of 7 items that are rated on a scale of 0 to 3. An overall Pittsburgh Sleep Quality Index score greater than 5 produced diagnostic sensitivity and specificity in distinguishing good and poor sleepers.
PSQI Change | Change from Baseline PSQI at 1 month
  It is a tool used to assess the quality of sleep in the last month.It consists of 7 items that are rated on a scale of 0 to 3. An overall Pittsburgh Sleep Quality Index score greater than 5 produced diagnostic sensitivity and specificity in distinguishing good and poor sleepers.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes M Fernández Seguín, PhD, Principal Investigator — University of Seville
Locations (1):
- Nursing, Physiotherapy and Podiatry Faculty, Seville, Spain, Spain